CLINICAL TRIAL: NCT00107523
Title: A Phase I Trial Evaluating the Effect of the Addition of HMGCoA-Reductase Inhibition With Pravastatin to Salvage Chemotherapy Idarubicin-HDAC in Patients With Relapsed or Refractory Acute Myelogenous Leukemia
Brief Title: Pravastatin, Idarubicin, and Cytarabine in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 1945.00; FHCRC-1945.00; MDA-2004-0185; CDR0000419678 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Pravastatin

INTERVENTIONS:
Drug: cytarabine
Drug: idarubicin
Drug: pravastatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Pravastatin may help idarubicin and cytarabine work better by making cancer cells more sensitive to the drugs. Giving pravastatin together with idarubicin and cytarabine may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of pravastatin when given together with idarubicin and cytarabine in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the biological efficacy of pravastatin in leukemia cells, in terms of measuring surrogate endpoints, including cellular cholesterol, messenger RNA encoding cholesterol synthesis, cholesterol import regulators, and specific protein farnesylation, in patients with acute myeloid leukemia.
* Determine whether increasing doses of pravastatin, when administered with idarubicin and high-dose cytarabine, produce increased apoptosis in leukemia cells of these patients.
* Determine the maximum tolerated dose (MTD) of pravastatin when administered with idarubicin and high-dose cytarabine in these patients.
* Determine whether the MTD of pravastatin is required to achieve the maximal biological effect on cholesterol metabolism in leukemia cells of these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of pravastatin.

Patients receive oral pravastatin once daily on days 1-8, idarubicin IV over 30 minutes on days 4-6, and high-dose cytarabine IV continuously on days 4-7. Treatment repeats every 28-42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete remission (CR) may receive additional treatment with the same doses of study drugs over fewer days. These patients receive oral pravastatin once daily on days 1-6 and idarubicin IV over 30 minutes and high-dose cytarabine IV continuously on days 4 and 5. Patients experiencing disease response with severe side effects may receive additional treatment at a lower dose of the study drug causing the side effects.

Cohorts of 3 patients receive escalating doses of pravastatin until the maximum tolerated dose (MTD)* is determined or a predetermined maximum dose is reached.

NOTE: *Patients achieving a CR with a dose of pravastatin that is subsequently determined to be above the MTD receive pravastatin at the MTD for all subsequent courses.

After completion of study treatment, patients are followed at least every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) meeting 1 of the following criteria:

  * Newly diagnosed disease (MDACC patients only)
  * In first or second relapse AND scheduled to receive first salvage therapy
  * Primary refractory disease after prior induction therapy for newly diagnosed disease

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* AST or ALT ≤ 2 times normal
* Alkaline phosphatase ≤ 2 times normal
* Bilirubin < 2.0 mg/dL
* No acute or chronic hepatic impairment

Renal

* Creatinine < 1.5 times normal (unless secondary to acute myeloid leukemia)

Cardiovascular

* Ejection fraction (EF) ≥ 45% by MUGA or 2-D echocardiogram

  * Patients who have an EF < 45% OR cardiac symptoms must be evaluated and cleared by cardiology to be eligible for study entry
* No cardiac contraindication to idarubicin

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled or life threatening infection
* No known intolerance to study drugs
* Must be able to safely tolerate the 3-day delay between the start of pravastatin and the start of chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent HMG-CoAR inhibitors, including any of the following:

  * Atorvastatin
  * Fluvastatin
  * Lovastatin
  * Rosuvastatin
  * Simvastatin
* No concurrent non-HMG-CoAR inhibitors to lower cholesterol
* No concurrent use of any of the following medications:

  * Bezafibrate
  * Clofibrate
  * Fenofibrate
  * Gemfibrozil
  * Cholestipol
  * Cholestyramine resin
  * Colesevelam
  * Ezetimibe
  * Biphenabid
  * Niacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Biological efficacy by measuring surrogate end-points, including cellular cholesterol, messenger RNAs encoding cholesterol synthesis and cholesterol import regulators, and specific protein farnesylation
Leukemia cell apoptosis
Maximum tolerated dose (MTD) of pravastatin
Maximal biological effect on cholesterol metabolism achieved with or without the MTD of pravastatin

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H. Petersdorf, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington